CLINICAL TRIAL: NCT01904890
Title: Asian American Network for Cancer Awareness, Research, and Training (AANCART): The National Center for Reducing Asian American Cancer Health Disparities Research Project on Lay Health Workers and Asian Americans
Brief Title: AANCART Research Project on Lay Health Workers and Asian Americans
Acronym: AANCARTLHW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); University of California, Los Angeles (Other); University of Hawaii (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U54CA153499 Sub7323; U54CA153499 (NIH)
Record Dates: First submitted 2013-07-10; First posted 2013-07-22 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: Asian Americans; colorectal cancer screening; cancer prevention; Filipinos Americans; Hmong Americans; Korean Americans; Randomized Controlled Trials
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRC Prevention and Screening Education (Experimental): Intervention Lay Health Workers (LHWs) will be taught to teach their participants about CRC screening through 2 outreach sessions and 2 telephone calls aimed at increasing their CRC screening receipt.
  Interventions: Behavioral: CRC Prevention and Screening Education
- Nutrition Education (Active Comparator): LHWs and participants in the comparison group will receive a bilingual CRC brochure as well as 2 lectures on healthy nutrition for cardiovascular health delivered by a health educator and an optional post- intervention LHW outreach session on CRC screening.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: CRC Prevention and Screening Education — Refer to Arm Description
  Arms: CRC Prevention and Screening Education
Behavioral: Nutrition Education — Refer to Arm Description
  Arms: Nutrition Education

SUMMARY:
This is a behavioral research study to evaluate the effectiveness of a type of health education, lay health worker (LHWs), on increasing the use of a routine health behavior, colorectal cancer (CRC) screening, among Asian Americans, who underutilize such screening. Using quantitative and qualitative methods and a community-based participatory research (CBPR) approach, the project will develop and implement a group randomized controlled trial to evaluate LHW effectiveness in promoting CRC screening among Asian Americans age 50 to 75. The investigators will conduct focus groups and individual interviews with community participants to revise training and survey materials developed in prior projects. The investigators will recruit LHWs to be randomly assigned to the intervention arm and to the comparison arm. The LHWs will each recruit 15 participants from their social network. Intervention LHWs will be taught to teach their participants about CRC screening through 2 outreach sessions and 2 telephone calls aimed at increasing their CRC screening receipt. LHWs and participants in the comparison group will receive a bilingual CRC brochure as well as 2 lectures on healthy nutrition for cardiovascular health delivered by a health educator and an optional post- intervention LHW outreach session on CRC screening. Effectiveness of the intervention will be measured by pre-intervention and post-intervention surveys of community participants' CRC screening behaviors. The investigators will also conduct ethnographic observations of LHWs and their participants during the small group sessions and post- intervention focus groups to understand how such a health education approach may work.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Filipino, Hmong, or Korean Americans
* age 50 to 75
* speak a language that the lay health worker (LHW) can speak such as Tagalog, Ilocano, Hmong, Korean, or English
* live in relevant area and intend to stay there for at least 12 months
* are willing to participate in a study about health behaviors involving nutrition or CRC screening.

Exclusion Criteria:

* personal history of CRC
* medical problems which may prevent them from attending 2 educational sessions

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Receipt of CRC Screening | Baseline to 6 months
  self-report of ever had fecal occult blood test (FOBT), sigmoidoscopy, or colonoscopy

SECONDARY OUTCOMES:
Up-to-date CRC screening receipt | Baseline to 6 months
  self-report of FOBT within 12 months, sigmoidoscopy within 5 years, or colonoscopy within 10 years
CRC screening Intention | Baseline to 6 months
  self-report of intending to obtain CRC screening in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tung Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of Hawai'i at Manoa, Honolulu, Hawaii